CLINICAL TRIAL: NCT07150104
Title: A Phase I/II, Randomized, Open-label Platform Study Utilizing a Master Protocol to Study Belantamab Mafodotin (GSK2857916) as Monotherapy and in Combination With Anti-Cancer Treatments in Participants With Relapsed/Refractory Multiple Myeloma (RRMM)-DREAMM5 - Sub-study 7 - Belantamab Mafodotin, Nirogacestat, Pomalidomide, and Dexamethasone in Combination
Brief Title: Sub-study of Belantamab Mafodotin (GSK2857916) as Monotherapy and in Combination With Nirogacestat, Pomalidomide, and Dexamethasone in Participants With RRMM
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 208887 Sub Study 7; 2023-509550-55-00 (EU CTIS Number)
Expanded Access: NCT03763370 (Available)
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: Belantamab Mafodotin; Nirogacestat; Pomalidomide; Dexamethasone; GSK2857916; Multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; nirogacestat; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belantamab mafodotin + Nirogacestat + Pomalidomide + Dexamethasone (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Nirogacestat; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Belantamab mafodotin — Belantamab mafodotin will be administered.
  Other Names: GSK2857916
Drug: Nirogacestat — Nirogacestat will be administered.
Drug: Pomalidomide — Pomalidomide will be administered.
Drug: Dexamethasone — Dexamethasone will be administered.

SUMMARY:
The primary purpose is to determine the safety and tolerability of belantamab mafodotin in combination with nirogacestat, pomalidomide, and dexamethasone and to establish the recommended Phase 2 dose for combination treatment to explore in the cohort expansion (CE) phase in participants with RRMM. This study is a sub study of the Master protocol (NCT04126200).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age inclusive or older, at the time of signing the informed consent.
* Participants must have histologically or cytologically confirmed diagnosis of Multiple Myeloma (MM), as defined by the IMWG.
* Participants having at least 3 prior lines of prior anti-myeloma treatments including an immunomodulating agent (IMID) a proteasome inhibitor (PI) and an anti-CD38 monoclonal antibody.
* Participants with a history of autologous stem cell transplant are eligible for study participation when, transplant was >100 days prior to study enrolment and with no active infection(s).
* Participants with Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, unless ECOG less than equal to (<=)2 is due solely to skeletal complications and/or skeletal pain due to MM.
* Participants with measurable disease defined as at least one of the following: Serum M-protein greater than equal to (>=)0.5 gram per deciliter (>=5 gram per liter) or Urine M-protein >=200 milligrams (mg) per 24 hours or Serum free light chain (FLC) assay: Involved FLC level >=10 mg per deciliter (>=100 mg per Liter) and an abnormal serum FLC ratio (<0.26 or >1.65).
* Participants who have tested positive for Hepatitis B core antibody (HBcAb) can be enrolled if the following criteria are met: Serology result HBcAb+, Hepatitis B surface antigen (HBsAg)-; HBV deoxyribonucleic acid (DNA) undetectable during screening.
* Participants who are currently receiving physiological doses oral steroids (<10 mg/day), inhaled steroids or ophthalmalogical steroids.
* Participants with platelets value for Adequate Organ System Function is ≥75 × 10^9/L.

Exclusion Criteria:

* Participants with current corneal epithelial disease except mild punctate keratopathy.
* Participants with evidence of cardiovascular risk.
* Participants with known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to belantamab mafodotin or any of the components of the study treatment. History of severe hypersensitivity to other mAb.
* Participants with active infection requiring antibiotic, antiviral, or antifungal treatment.
* Participants with other monoclonal antibodies within 30 days or systemic anti-myeloma therapy within <14 days.
* Participants with prior radiotherapy within 2 weeks of start of study therapy.
* Participants with prior allogeneic transplant are prohibited.
* Participants who have received prior Chimeric Antigen T cell therapy (CAR-T) therapy with lymphodepletion with chemotherapy within 3 months of screening.
* Participants with any major surgery (other than bone-stabilizing surgery) within the last 30 days.
* Participants with prior treatment with an investigational agent within 14 days or 5 half-lives of receiving the first dose of study drugs, whichever is shorter.
* Participants with >=grade 3 toxicity considered related to prior check-point inhibitors and that led to treatment discontinuation.
* Participants who have received transfusion of blood products within 2 weeks before the first dose of study drug.
* Participants must not receive live attenuated vaccines within 30 days prior to first dose of study treatment or whilst receiving belantamab mafodotin +- partner agent in any sub-study arm of the platform trial and for at least 70 days following last study treatment.
* Participants with presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM.
* Participants with known human immunodeficiency virus (HIV) infection, unless the participant can meet all criteria: a) established anti-retroviral therapy for at least 4 weeks and HIV viral load<400 copies/milliliter (mL) b) cluster of differentiation 4 plus (CD4+) T-cell (CD4+) counts >= 350 cells/microliter (µL) c) No history of Acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections within the last 12 months in which case the participant would be eligible for CE Phase only. For participants receiving nirogacestat, HIV drugs that are strong Cytochrome P450 3A4 (CYP3A4) inhibitors are prohibited. HIV drugs that are moderate CYP3A4 inhibitors, while permitted, should be co-administered with caution and must be accompanied by nirogacestat dose modifications.
* Participants with uncontrolled small and/or large intestinal disease.
* Participants with uncontrolled skin disease.
* Participants with any condition causing hypophosphatemia, hypokalemia or hypomagnesemia which is refractory to electrolyte replacement.
* Participants with previous administration of a gamma secretase inhibitor.
* Participants with concomitant administration of a strong CYP3A4 inhibitor or inducer.
* Participants with active or history of venous thromboembolism within the past 3 months.
* Participants with evidence of active mucosal or internal bleeding.
* Participants with contraindications to or are unwilling to undergo protocol-required anti-thrombotic prophylaxis or unable to tolerate antithrombotic prophylaxis.
* Participants who discontinued prior treatment with pomalidomide due to intolerable adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2027-03-11 (Estimated)

PRIMARY OUTCOMES:
Dose Exploration (DE) Phase: Number of participants with dose limiting toxicities (DLTs) | Up to 21 days
DE Phase: Number of participants with adverse events (AEs) | Up to approximately 137 weeks
DE Phase: Number of participants with clinically significant changes in hematology, clinical chemistry, and urinalysis lab parameters | Up to approximately 137 weeks
Cohort Expansion (CE) Phase: Overall Response Rate (ORR) | Up to approximately 137 weeks
  ORR is defined as the percentage of participants with a confirmed Partial response (PR) or better as the best overall response (BOR), according to the International Myeloma Working Group (IMWG) Response Criteria.

SECONDARY OUTCOMES:
DE Phase: Overall Response Rate | Up to approximately 236 weeks
  ORR is defined as the percentage of participants with confirmed PR or better as BOR, according to the IMWG Response Criteria.
CE Phase: Clinical Benefit Rate (CBR) | Up to approximately 236 weeks
  CBR is defined as the percentage of participants with a confirmed minimal response (MR) or better as BOR, according to IMWG response criteria.
DE Phase: Number of participants achieving Partial Response (PR) | Up to approximately 236 weeks
  Number of participants with PR according to IMWG criteria will be analysed.
CE Phase: Number of participants achieving PR | Up to approximately 236 weeks
  Number of participants with PR according to IMWG criteria will be analysed.
DE Phase: Number of participants achieving Very Good Partial Response (VGPR) | Up to approximately 236 weeks
  Number of participants with VGPR according to IMWG criteria will be analysed.
CE Phase: Number of participants achieving VGPR | Up to approximately 236 weeks
  Number of participants with VGPR according to IMWG criteria will be analysed.
DE Phase: Number of participants achieving Complete Response (CR) | Up to approximately 236 weeks
  Participants with CR according to IMWG criteria will be analysed.
CE Phase: Number of participants achieving CR | Up to approximately 236 weeks
  Participants with CR according to IMWG criteria will be analysed.
DE Phase: Number of participants achieving Stringent Complete Response (sCR) | Up to approximately 236 weeks
  Participants with sCR according to IMWG criteria will be analysed.
CE Phase: Number of participants achieving sCR | Up to approximately 236 weeks
  Participants with sCR according to IMWG criteria will be analysed.
DE Phase: Belantamab mafodotin concentrations when administered in combination with anti-cancer treatments | Up to approximately 236 weeks
CE Phase: Belantamab mafodotin concentrations when administered in combination with anti-cancer treatments | Up to approximately 236 weeks
DE Phase: Nirogacestat concentration when administered in combination with belantamab mafodotin | Up to approximately 236 weeks
CE Phase: Nirogacestat concentration when administered in combination with belantamab mafodotin | Up to approximately 236 weeks
DE Phase: Pomalidomide concentration when administered in combination with belantamab mafodotin | Up to approximately 236 weeks
CE Phase: Pomalidomide concentration when administered in combination with belantamab mafodotin | Up to approximately 236 weeks
DE Phase: Dexamethasone concentration when administered in combination with belantamab mafodotin | Up to approximately 236 weeks
CE Phase: Dexamethsone concentration when administered in combination with belantamab mafodotin | Up to approximately 236 weeks
DE Phase: Number of participants with anti-drug antibodies (ADAs) against belantamab mafodotin | Up to approximately 236 weeks
DE Phase: Titre of (ADAs) against belantamab mafodotin | Up to approximately 236 weeks
CE Phase: Number of participants with ADAs against belantamab mafodotin | Up to approximately 236 weeks
CE Phase: Titre of ADAs against belantamab mafodotin | Up to approximately 236 weeks
DE Phase: Number of participants with adverse events of special interest (AESI) for belantamab mafodotin | Up to approximately 236 weeks
CE Phase: Number of participants with AESI for belantamab mafodotin | Up to approximately 236 weeks
DE Phase: Number of participants with AESI for Nirogacestat | Up to approximately 236 weeks
CE Phase: Number of participants with AESI for Nirogacestat | Up to approximately 236 weeks
DE Phase: Number of participants with AESI for Pomalidomide | Up to approximately 236 weeks
CE Phase: Number of participants with AESI for Pomalidomide | Up to approximately 236 weeks
DE Phase: Number of participants with AESI for Dexamethasone | Up to approximately 236 weeks
CE Phase: Number of participants with AESI for Dexamethasone | Up to approximately 236 weeks
DE Phase: Number of participants with abnormal ocular findings on ophthalmic examination | Up to approximately 236 weeks
CE Phase: Number of participants with abnormal ocular findings on ophthalmic examination | Up to approximately 236 weeks
CE Phase: Progression-free survival (PFS) | Up to approximately 236 weeks
  PFS is defined as the time from randomization until the earliest date of confirmed progressive disease (PD) per IMWG, or death due to any cause.
CE Phase: Duration of response (DoR) | Up to approximately 236 weeks
  DoR is defined as the time from first documented evidence of confirmed PR or better until progressive disease per IMWG or death due to progressive disease among participants who achieve confirmed partial response or better.
CE Phase: Time to response (TTR) | Up to approximately 236 weeks
  TTR is defined as the time between the date of randomization and the first documented evidence of response (confirmed PR or better), among participants who achieve a response (confirmed PR or better).
CE Phase: Overall survival (OS) | Up to approximately 236 weeks
  OS is defined as the time from randomization until death due to any cause.
CE Phase: Number of participants with AEs and SAEs | Up to approximately 236 weeks
CE Phase: Number of participants with AEs leading to discontinuation | Up to approximately 236 weeks
CE Phase: Number of participants with AE leading to dose reduction or delay | Up to approximately 236 weeks
CE Phase: Number of participants with clinically significant changes in hematology, clinical chemistry and urinalysis lab parameters | Up to approximately 236 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- Brazil (2):
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
- GSK Investigational Site, Halifax, Nova Scotia, Canada
- GSK Investigational Site, Villejuif, France
- GSK Investigational Site, Mexico City, Mexico
- GSK Investigational Site, Oslo, Norway
- GSK Investigational Site, Lublin, Poland
- South Korea (2):
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Ulsan
- GSK Investigational Site, Falun, Sweden

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.